CLINICAL TRIAL: NCT05710536
Title: Safety and Efficacy of Formulation Containing Stem Cell Secretome and Liquorice Root Extract for Improving Vagina Laxity of Women in Malaysia: A Pilot Study.
Brief Title: Safety and Efficacy of Formulation for Improving Vagina Laxity: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UMRAMREC006-22
Record Dates: First submitted 2023-01-13; First posted 2023-02-02 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: Vagina laxity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Formulation X (Experimental): Participants will use the formulation once every 72 hour for 5 weeks
  Interventions: Other: Formulation X

INTERVENTIONS:
Other: Formulation X — This formulation containing stem cell secretome and liquorice root extract

SUMMARY:
This study is conducted to investigate the safety and efficacy of the formulation containing stem cell secretome and licorice root extract in improving vagina laxity (VL) condition of women in Malaysia. This formulation may stimulate cell rejuvenation and trigger cell renewal efficiently as they contained rich mixture of natural, bioavailable polypeptides and plant extracts and these might help improving the VL condition in women. The study duration is 5 weeks and vagina assessment will be carried out at baseline, week 2 and week 5.The main objectives of this study are:

1. To assess the vagina laxity of women in Malaysia after using the formulation.
2. To observe any adverse effect occurrence with the use of the formulation.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian women ( age 40 to 55 years old)
* Complaint of vagina laxity
* Willingness to participate in the study

Exclusion Criteria:

* Pregnant and breastfeeding women
* Doing any surgical or non-surgical procedures to improved vaginal laxity condition such as laser and radiofrequency before participating in the study that might affect the study outcome
* Presence of illness or taking any medication that might impact the study outcome or participants well-being

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 18 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in vagina laxity condition from baseline and at week 2 and week 5 after using the product | Baseline, Week 2 and Week 5
  Vagina laxity questionnaire (VLQ) will be used to assess participant's vagina laxity conditions at baseline, week 2 and week 5. This is a self-reported tool where participants will be asking to score their vagina laxity on a scale of 1 to 7 (1= very loose, 2= moderately loose, 3= slightly loose, 4= neither tight nor loose, 5= very tight, 6= moderately tight, 7= very tight)
Change in vagina tone from baseline and at week 2 and week 5 after using the product | Baseline, Week 2 and Week 5
  Vagina tone is measured using a perineometer (measurement of vaginal squeeze pressure). This assessment will be carried out by trained clinician at baseline, week 2 and week 5 and it will determine participant vagina tone.
Adverse effect after using the formulation | week 5
  Based on adverse effect occurrence on participants that occur during study period (5 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No